CLINICAL TRIAL: NCT04825496
Title: Clinical Study of ssCART-19 Cells in Patients With CD19 Positive Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ssCART-19
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-05

CONDITIONS: Relapsed or Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ssCART-19 Cells (Experimental): Route of administration: Intravenous injection.
  Lymphodepletion conditioning:
  Lymphodepletion will be conducted several days prior to ssCART-19 cells infusion.
  A combination of fludarabine and cyclophosphamide will be used for lymphodepletion.
  Interventions: Genetic: ssCART-19 Cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: ssCART-19 Cells — Split-Dose of ssCART-19 cells will be infused, and classic "3+3" dose escalation will be applied.
Drug: Fludarabine — Fludarabine is used for lymphodepletion.
  Other Names: FA
Drug: Cyclophosphamide — Cyclophosphamide is used for lymphodepletion.
  Other Names: CTX

SUMMARY:
This is a single arm, open-label, non-randomized, dose-escalation, phase I study to determine the safety and efficacy of ssCART-19 in the treatment of patients with CD19 positive relapsed or refractory acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
This is a single arm, open-label, non-randomized, dose-escalation, phase I study to determine the safety and efficacy of ssCART-19 in the treatment of patients with CD19 positive relapsed or refractory acute lymphoblastic leukemia.

Primary objectives:

Determine the safety and tolerability of ssCART-19 cells in patients with refractory or relapsed acute lymphoblastic leukemia.

Secondary objectives:

1. Observe the anti-tumor response of ssCART-19 cells to refractory or relapsed acute lymphoblastic leukemia.

   * Overall remission rate (ORR) assessment during the 3 months after ssCART-19 administration，ORR includes CR and CRi
   * Duration of response (DOR)
   * Progression-free survival (PFS)
   * Overall survival (OS)
2. To characterize the in vivo cellular pharmacokinetic (PK) profile of ssCART-19 cells.
3. To characterize the pharmacodynamic (PD) profile of ssCART-19 cells.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory acute lymphoblastic leukemia (ALL):(1)Any Relaps after first remission OR (2)Any BM relapse after allogeneic SCT and must be ≥ 3 months from SCT at the time of ssCART-19 infusion OR (3)failed to reach CR after 2 cycles of induction chemotherapy regimen OR (4)Patients with Ph+ ALL are eligible if they are intolerant to or have failed two lines of TKI therapy, or if TKI therapy is contraindicated
2. CD19 tumor expression demonstrated in bone marrow or peripheral blood by flow cytometry
3. Bone marrow with ≥ 5% lymphoblasts by morphologic assessment
4. Adequate organ function defined as:(1)left ventricular ejection fraction ≥ 50% by echocardiogram；(2)creatinine ≤ 1.6mg/dl；(3)ALT and AST≤3 times the ULN for age, total bilirubin ≤ 2.0mg/dl；(4)Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygenation > 91% on room air
5. Informed consent is signed by the subject
6. Age 18 to 65
7. Fertility of men, to ensure that sexual partners can effectively contraception; Women with fertility use effective contraceptive measures and agree to use contraceptive measures throughout the study period
8. Qualified T cell amplification
9. Eastern cooperative oncology group (ECOG) performance status of 0 to 1
10. Vascular conditions for apheresis
11. The estimated survival time is more than 3 months

Exclusion Criteria:

1. Isolated extra-medullary disease relapse
2. Combined with other malignant tumors
3. Has had treatment with any prior anti-CD19/anti-CD3 therapy, or any other antiCD19 therapy
4. Has had immunosuppressants or hormones within 2 weeks before signing informed consent, or plan to use immunosuppressants or hormones after signing informed consent
5. Patients complying with any of hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg) positive, hepatitis B e antibody (HBe-Ab) and/or hepatitis B core antibody (HBc-Ab) positive and HBV-DNA copies being more than the lower limit of detection, hepatitis C antibody (HCV-Ab) positive, anti-treponemia pallidum antibody (TP-Ab) positive, EBV-DNA, and CMV-DNA copies being more than the lower limit of detection
6. Has uncontrolled bacteria, fungi, viruses, mycoplasma or other types of infections
7. Infected with HIV, syphilis or COVID-19
8. Has a history of severe immediate hypersensitivity to aminoglycosides
9. Has past or present CNS diseases, such as epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar diseases or any CNS-related autoimmune diseases
10. Has undergone cardiac angioplasty or stent implantation within 12 months before signing informed consent, or having a history of myocardial infarction, unstable angina pectoris or other clinically significant heart diseases
11. With primary immunodeficiency
12. Has had severe immediate hypersensitivity reaction to any drug to be used in this study
13. Has had treat with live vaccine within 6 weeks prior to screening
14. Pregnant or lactating women
15. Has active autoimmune diseases
16. Has active acute or chronic graft-versus-host disease (GVHD) before signing informed consent
17. Patient has an investigational medicinal product within 3 months before signing informed consent
18. Patients with other conditions making the patients unsuitable for receiving cell therapy as judged by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 28 days
  Determine the safety and tolerability of ssCART-19 in patients with refractory or relapsed acute lymphoblastic leukemia.
  Safety measures include adverse events as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Overall Remission Rate (ORR), which includes Complete Remission (CR) and Complete Remission with Incomplete Blood Count Recovery (CRi) | 3 months
  Efficacy of ssCART-19 as measured by ORR during the 3 months after ssCART-19 infusion, which includes CR and CRi.
Duration of remission (DOR) | 24 months
  Statistical parameter:Duration of remission (DOR)
Progression-free Survival (PFS) | 24 months
  Statistical parameter:Progression-free Survival (PFS)
Overall survival (OS) | 24 months
  Statistical parameter:Overall survival (OS)

OTHER OUTCOMES:
cellular pharmacokinetic (PK) profile of ssCART-19 cells | 24 months
  Number of DNA copies of ssCART-19 cells
Anti-drug antibody | 24 months
  Detect titer of anti-drug antibody (ADA)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Unicar-Therapy Bio-medicine Technology Co., Ltd., Shanghai, Shanghai Municipality, China